CLINICAL TRIAL: NCT00380224
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group Fixed-Dose Study of the Effect on Weight of Befeprunox Versus Olanzapine in the Treatment of Outpatients With Schizophrenia.
Brief Title: Study Comparing the Affect of Bifeprunox Vs Olanzapine on Weight During the Treatment of Outpatients With Schizophrenia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3168A1-311
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Schizophrenia
Keywords: schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — bifeprunox; Olanzapine

INTERVENTIONS:
Drug: bifeprunox, olanzapine

SUMMARY:
This study will compare bifeprunox to a currently marketed medication, Zyprexa (olanzapine), with respect to the affect on weight during the treatment of outpatients with schizophrenia. The study will compare the effect of these medications on several variables, including body weight and triglyceride levels.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel-group study of bifeprunox in the treatment of outpatients with schizophrenia, with olanzapine as the active comparator. Subjects must be stable for 3 months or more of treatment with olanzapine at baseline. There will be 2 treatment arms in this study, approximately 60 subjects per arm. After randomization and blinding, each subject will either remain on olanzapine or switch to bifeprunox. Assessments, including body weight and waist measurements, will be made at each study visit.Subjects will participate in the study for approximately 11 weeks. After a screening period of 6 to 14 days, eligible subjects will be treated for 8 weeks. Subjects who do not enter the long-term extension will return for a follow-up visit 7 days after discontinuing the use of test article. Subjects who do enter the long-term extension will have a 7-day taper/titration period after the 8 weeks of double-blind treatment.

ELIGIBILITY:
Inclusion criteria:

* Current treatment of at least 3 months with olanzapine.
* Primary diagnosis of schizophrenia.
* Total Positive and Negative Symptoms Scale (PANSS) score <=70 at screening and baseline.

Exclusion criteria:

* Psychiatric diagnosis other than schizophrenia, as assessed by the modified Mini International Neuropsychiatric Interview (MINI), and considered by the investigator to be the primary psychiatric diagnosis.
* History or presence of clinically significant cardiovascular, endocrine, hepatic, renal or other medical disease that might be detrimental to the subject or confound the study.
* History of any suicide attempt within 3 years of day -1 or significant immediate risk of violence or suicidality.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-07; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline on body weight at the final evaluation.

SECONDARY OUTCOMES:
Change from baseline in triglyceride level; Change from baseline in waist circumference; and Change from baseline in total Positive and Negative Syndrome Scale (PANSS) score.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (58):
- United States (58):
  - Little Rock, Arkansas
  - Anaheim, California
  - Boynton Beach, California
  - Costa Mesa, California
  - Escondido, California
  - Garden Grove, California
  - Glendale, California
  - Huntington Beach, California
  - La Mesa, California
  - National City, California
  - Oceanside, California
  - Paramount, California
  - Rosemead, California
  - San Diego, California
  - Santa Ana, California
  - New Britain, Connecticut
  - New London, Connecticut
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - North Miami, Florida
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Marietta, Georgia
  - Coevr d'Alene, Idaho
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Joliet, Illinois
  - Naperville, Illinois
  - Lake Charles, Louisiana
  - Gaithersburg, Maryland
  - Worcester, Massachusetts
  - Flowood, Mississippi
  - St Louis, Missouri
  - North Platte, Nebraska
  - Cherry Hill, New Jersey
  - Clementon, New Jersey
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - Butner, North Carolina
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Morehead City, North Carolina
  - Fargo, North Dakota
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Norristown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Cordova, Tennessee
  - Memphis, Tennessee
  - Murfressboro, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - DeSoto, Texas
  - Irving, Texas